CLINICAL TRIAL: NCT03359941
Title: Acupuncture Treatment for Pain Relief and Functional Recovery in Patients With Vertebral Compression Fracture
Brief Title: Acupuncture Treatment for Vertebral Compression Fracture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruit rate
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N2015002
Record Dates: First submitted 2015-12-10; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Spinal Fracture; Compression Fracture; Fractures, Bone
Keywords: Integrative Treatments; Korean Traditional medicine
MeSH Terms: conditions — Spinal Fractures; Fractures, Compression; Fractures, Bone | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Integrative Treatments (Experimental): This study's arm is single, so all participants will receive acupuncture treatments.
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — Acupuncture points: Examples of acupuncture points to be used include BL23 (Sinsu, bilateral), BL24(Gihaesu, bilateral), BL25(Daejangsu, bilateral), BL40(Wijung, bilateral), BL60(Gollyun, bilateral), BL65(Sokgol, bilateral), LI11(Gokji, bilateral), LI4(Hapgok, bilateral), ST36(Joksamni, bilateral), GB41(Jogimeup, bilateral), LR3(Taechung, bilateral). Electrical stimulation with alternating frequency of 2-100 Hz will be applied to the selected points (e.g., BL 23-25, bilateral). Treatments will be provided by qualified Korean traditional medicine doctors with more than 2 years of clinical experience.

SUMMARY:
Patients with vertebral compression fractures (VCF) may experience pain, limitation of daily activities, and various complications (e.g., insomnia, constipation, urinary infection, depression, diminished quality of life).

Objective:

This study aims to evaluate the effectiveness, safety and feasibility of acupuncture treatments to achieve pain relief and functional recovery in patients with VCF.

DETAILED DESCRIPTION:
Patients who have subacute or chronic vertebral compression fracture in one or more thoracic/lumbar vertebral body are eligible. Patients who have willingness to participate and provide written informed consents will be treated to the Pusan National University Korean Medicine Hospital with once to three times per weak for six weeks approximately. (total 12-18 sessions)

ELIGIBILITY:
Inclusion Criteria:

* Is at least 19 years of age
* Radiographic confirmation of one more subacute or chronic stable vertebral compression fractures (x-ray, computerized tomography, or magnetic resonance imaging)
* Patient-reported pain intensity equal or greater than 4 points on 0 to 10 VAS scale at baseline
* Willingness to participate in the study and provide written informed consent
* Is able to give written consent independently or with a supporter's help

Exclusion Criteria:

* Pathological fracture (malignancy, myeloma, metabolic disease, etc.)
* Spine malformation
* Pregnancy, infection, impaired cognitive function
* Hypersensitive reaction to acupuncture treatment
* Need for surgical treatment

  1. Neurologic deficit: spinal cord injury, cauda equina syndrome
  2. Unstable fracture: three-column collapse, burst fracture, posterior ligament rupture, distraction fracture
  3. Scoliotic angle ≥ 12°

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Pain intensity on the Visual Analog Scale (VAS) | 6 weeks from the first treatment
  VAS will be used to assess pain intensity reflecting average patient-perceived pain during the previous 24 hours. The scale ranges from 0 (no pain) to 10 (the worst pain imaginable).

SECONDARY OUTCOMES:
Patient's satisfaction with treatment using the Patient Global Assessment(PGA) | 6 weeks from the first treatment
  Response options include very much satisfied, somewhat satisfied, neutral, somewhat dissatisfied, and very much dissatisfied.
Back-specific dysfunction using the Oswestry Disability Index (ODI) | baseline, 6 weeks from the first treatment, 12 weeks from the first treatment
  The questionnaire has 10 items to assess limitations of various activities of daily living. Each section is scored on a 0-5 score. Total scores are reported from 0 to 100, with higher scores indicating greater disability.
Quality of life using the Quality-of-Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO) | baseline, 6 weeks from the first treatment, 12 weeks from the first treatment
  QUALEFFO is used to evaluate the effect of back pain and treatment on quality of life. The questionnaire includes 26 items in 5 domains; pain, physical function, social function, general health perception, and mental function. Total scores are reported from 0 to 100, with lower scores corresponding to better quality of life.
Physical function using Time Up and Go (TUG) | baseline, 6 weeks from the first treatment
  TUG measures the time taken to stand from a chair, walk 3 meters, turn, and return to sitting in the chair.
Adverse events related to integrative treatments as a measure of safety | under treatment, 6 weeks from the first treatment, 12 weeks from the first treatment
  Expected or unexpected adverse events will be measured during the allocated intervention process and during the entire follow-up period. Both the types of adverse events and their frequency of occurrence will be measured.
Use of medication for pain control during treatment | under treatment, 6 weeks from the first treatment, 12 weeks from the first treatment
  Information on the use of medication will be collected by directly asking the patient at every visit. Medication type, dose, and frequency will be recorded and assessed.
Number of patients who received surgery | 12 weeks from the first treatment
  The number of patients who participated in the trial but finally received surgery during the study period will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Hyung Kim, PhD, Principal Investigator — Korean Medicine Hospital of Pusan National University
Locations (1):
- National Clinical Research Centre for Korean Medicine, Korean Medicine Hospital, Pusan National University, Yangsan, Kyung Sang South Province, South Korea

IPD SHARING:
Plan to Share IPD: No